CLINICAL TRIAL: NCT07077278
Title: Effect of Low Sodium Oxybate (LXB) on Autonomic Symptom Burden in Idiopathic Hypersomnia Patients With Postural Tachycardia Syndrome: a Placebo-controlled, Double-blind, Randomized Withdrawal Study
Brief Title: Effect of Low Sodium Oxybate (LXB) on Autonomic Symptom Burden in Idiopathic Hypersomnia Patients With Postural Tachycardia Syndrome
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Mitchell Miglis, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 75300
Record Dates: First submitted 2025-07-11; First posted 2025-07-22 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Hypersomnia; POTS - Postural Orthostatic Tachycardia Syndrome
MeSH Terms: conditions — Idiopathic Hypersomnia; Postural Orthostatic Tachycardia Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low sodium oxybate (LXB) (Experimental): Participants will take LXB for two weeks.
  Interventions: Drug: Low sodium oxybate (LXB)
- Placebo (Placebo Comparator): Participants will take placebo for two weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low sodium oxybate (LXB) — Participants will continue take low sodium oxybate (LXB) for two weeks after completing an open-label titration and dose optimization period of low sodium oxybate (LXB).
  Arms: Low sodium oxybate (LXB)
Drug: Placebo — Participants will take placebo for two weeks after completing an open-label titration and dose optimization period of low sodium oxybate (LXB).
  Arms: Placebo

SUMMARY:
The investigators hope to learn if low sodium oxybate (LXB) is an effective treatment for symptoms of idiopathic hypersomnia (IH) and postural tachycardia syndrome (POTS). Previous research has shown that patients with IH also report having symptoms associated with POTS. The researchers have observed that in patients with both IH and POTS, when patients' sleep quality improves, so do their POTS symptoms. The goal of this study is to test this in a controlled way by using LXB as a treatment for both IH and POTS in patients that have been diagnosed with both conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. English speaking and capable of signing the informed consent form and comply with the protocol requirements
3. Diagnosis of IH based on ICSD-3 criteria
4. Diagnosis of POTS based on the 2011 Consensus Criteria
5. Oxybate naïve. Participants on daytime alerting medications at baseline can remain on these medications for the duration of the study, provided doses remain stable for the duration of the study. This rule also applies to medications prescribed for the treatment of POTS. All medications known to affect cardiovascular function will be held for the appropriate time periods prior to active stand testing so as not to influence results.
6. COMPASS 31 ≥ 40 at the screening visit
7. Agree to use contraceptives consistent with local regulations regarding the methods of contraception for those participating in clinical trials

Exclusion Criteria:

1. Hypersomnia due to another medical, behavioral, sleep, or psychiatric disorder
2. Evidence of untreated or inadequately treated sleep disordered breathing, defined as AHI ≥ 10
3. History of bipolar or psychotic disorders, major depressive episode, or current suicidal risk
4. Pregnant or lactating or intends to become pregnant during the study
5. History of or currently being treated for clinically significant ongoing cardiac arrythmia, heart failure, myocarditis, pulmonary embolism requiring anticoagulation, pulmonary fibrosis or other pulmonary diagnosis that in the investigator's opinion may contribute to symptoms of POTS
6. Clinically significant uncontrolled active or chronic bacterial, viral, or fungal infection or positive SARS-CoV-2 PCR test at screening
7. A medical condition that could confound the results of the study or put the participant at undue risk in the investigator's judgment
8. Intends to have surgery or procedures requiring anesthesia or conscious sedation during the study
9. Currently participating in another interventional clinical study
10. Unwilling to remain on a stable regimen of medications during the study
11. Use of or planned use of intravenous saline infusions during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Overall COMPASS-31 Score as a measure of direct comparison between the two conditions across the two-week randomized withdrawal period. | At the end of the two-week randomized withdrawal period
  The Composite Autonomic Symptom Severity Scale-31 (COMPASS-31) is an overall assessment of autonomic symptom severity. The scale measures neurodegenerative system symptoms through 31 patient-reported questions. Assessment is through six weighted domains: orthostatic intolerance [10 points]; vasomotor [6 points]; secretomotor [7 points]; gastrointestinal [28 points]; bladder [9 points] and pupillomotor [15 points]. Weighted scores are summed. A higher score indicates worse autonomic dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Miglis, MD, Principal Investigator — Stanford University